CLINICAL TRIAL: NCT02328950
Title: A 5 Day Course of Fludarabine and Cytarabine Followed by Full Intensity Allogeneic Stem Cell Transplantation (FA5-Bucy) in Treating Patients With High-risk, Recurrent or Refractory Acute Leukemia and Advanced Myelodysplastic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ting YANG, Prof. Dr., Fujian Medical University
Other Study IDs: FA5Bucy-SCT-01
Record Dates: First submitted 2014-12-28; First posted 2014-12-31 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fludarabine and Cytarabine followed by IV busulfan and cyclophosphamide — Fludarabine (F) 30 mg/m²/day for 5 days (day -12 to day-8) Cytarabine (A) 2g/m²/day for 5 days (day -12 to day-8) Bulsufan (Bu) 0.8mg/kg/day for 3 days (day -7 to day-5) Cyclophosphamide(Cy) 1.8g/m²/day for 3 days (day -4 to day-3)

SUMMARY:
A 5 day course of fludarabine and cytarabine (FA) will be administered followed by full intensity conditioning regimen (Bucy) in the setting of allogeneic stem cell transplantation (SCT). The purpose of this study is to explore the antileukemic, immunosuppressive effects and safety of FA as the backbone of a conditioning regiment for the treatment of patients with high-risk, recurrent or refractory acute Leukemia and advanced myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Aged between 0-65 years
* Patients suffering from either refractory de novo AML/ALL or relapsed AML/ALL or patients with very high risk AML/ALL in CR1
* Patients with advanced MDS
* Cardiac: Left ventricular ejection fraction ≥ 50%
* Adequate renal and hepatic function
* Performance status: Karnofsky ≥ 70%

Exclusion Criteria:

* Pregnant or lactating females
* Current participation in another clinical trial
* Contra-indication to one of the drug of the regimen
* Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo the agents included in the conditioning regimen

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with high-risk, recurrent or refractory acute leukemia and advanced myelodysplastic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Relapse rate at one year after allo-SCT | one year

SECONDARY OUTCOMES:
Even free survival | two year
  * Overall Survival
  * Leukemia Free Survival
  * Graft Versus Host Disease
  * Regimen related toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital,Fujian Medical University, Fuzhou, Fujian, China